CLINICAL TRIAL: NCT02474901
Title: Shedding, Immunogenicity and Safety of Quadrivalent Live Intranasal Influenza Vaccine (QLAIV) in HIV-infected Children and Young Adults
Acronym: QLAIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-1752
Record Dates: First submitted 2015-06-15; First posted 2015-06-18 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Shedding; Immunogenicity; Safety; HIV infected; Children; Young adults
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QLAIV, HIV-infected (Active Comparator): QLAIV administered to HIV-infected individuals 2 to 25 yoa
  Interventions: Biological: Quadrivalent Live Attenuated Influenza Vaccine
- QLAIV, HIV-uninfected (Active Comparator): QLAIV administered to HIV-uninfected individuals 2 to 25 yoa
  Interventions: Biological: Quadrivalent Live Attenuated Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Live Attenuated Influenza Vaccine
  Other Names: FluMist Quadrivalent; QLAIV

SUMMARY:
The goal of this study is to determine if there is a difference in shedding (primary objective) and in immunogenicity and safety (secondary objectives) between HIV-positive and HIV-negative children and young adults who are receiving the quadrivalent live-attenuated influenza vaccine (QLAIV).

DETAILED DESCRIPTION:
QLAIV is an intranasal vaccine that works by using 4 different attenuated strains of influenza virus that will replicate in the nose and stimulate an immune response in recipients that should protect them if they are infected with one of those strains of influenza in the future. A couple of studies have shown an increase in duration that the viruses remain in the nose in immunocompromised people. Those studies were done using the trivalent vaccine, so the investigators would like to evaluate the quadrivalent vaccine, and there is still a need for additional data to help understand the duration of shedding. If shedding is prolonged in HIV-infected children and young adults, it would be important to know for contacts of those individuals who are very immunocompromised. Shedding will be measured by looking for influenza RNA in nasopharyngeal swabs taken at baseline, 2-5 days, 7-10 days and 14-21 days after the intranasal immunization.

The live-attenuated influenza vaccines have been shown to have increased effectiveness in children and they stimulate the immune system in a different way than the inactivated influenza vaccines (TIV or QIV). In this study, the investigators will have the opportunity to compare the immunogenicity of QLAIV, measured at baseline and 14-21 days post-vaccination, in HIV-infected and uninfected children, adolescents and young adults. Although prior studies of LAIV in HIV-infected and other immunocompromised children and adults have not shown any increase in serious adverse events, safety will be actively monitored for the first 30-45 days through a study-specific questionnaire administered at each clinic or phone visit and by asking the subjects to keep a diary of side effects. Safety will be monitored passively throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-25
* Only supposed to get one dose of vaccine for upcoming influenza season
* No viral respiratory symptoms at time of immunization
* HIV-infected group: must have:

  * HIV-infection documented by 2 tests such as positive serology, positive HIV DNA or positive HIV RNA;
  * must thave a CD4>25% or 500, or
  * must have CD4>15% or 200 and be on HAART
* Healthy controls: no major medical problems affecting the immune system
* Recruited among:

  * HIV-unifected clients of the Children's Immunodeficiency Program(CHIP),
  * Children's Hospital Colorado Child Health Clinic and Adolescent Clinics.

Exclusion Criteria:

* History of:

  * reactive airway disease,
  * recurrent wheezing, or
  * asthma
* Active wheezing at time of immunization
* On any antiviral agents active against influenza (amantadien/rimantadine, zanamavir, oseltamivir) at time of immunization or planned over 21 days of shedding collection
* Receipt of IVIG within 3 months prior to enrollment
* Plan to receive IVIG during the 4 weeks after immunization
* Moderate to severely immunocompromised individual living in the home
* Pregnant
* Breastfeeding
* Plan to start immunosupressive medications or stop HAART over the 4 weeks following immmunization
* Temperature > 100F or 37.8C
* Rhinorrhea or cough not related to allergies at the time of immunization
* History of fungal sinusitis
* History of Guillain-Barre Syndrome
* Current on antibiotics
* Currently taking aspirin
* On an investigational drug at the time of immunization or planned over the 28 days of shedding collection
* On any experimental medication at time of immunization or planned over 21 days of shedding collection

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Weinberg, MD, Principal Investigator — University of Colorado, Denver; Myron Levin, MD, Study Chair — University of Colorado, Denver; Donna Curtis, MD,MPH, Study Director — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- QLAIV, HIV-uninfected: QLAIV administered to HIV-uninfected individuals 2 to 25 yoa
  Quadrivalent Live Attenuated Influenza Vaccine
- QLAIV, HIV-infected: QLAIV administered to HIV-infected individuals 2 to 25 yoa
  Quadrivalent Live Attenuated Influenza Vaccine
Period: Overall Study
Arm/Group | QLAIV, HIV-uninfected | QLAIV, HIV-infected
Started | 45 | 56
Completed | 44 | 56
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QLAIV, HIV-infected | QLAIV, HIV-uninfected | Total
Number analyzed (Participants) | 45 | 56 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 22 | 32
  Between 18 and 65 years | 35 | 34 | 69
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 18 [10 to 23] | 10 [7 to 14] | 12 [8 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 26 | 43
  Male | 28 | 30 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 13 | 20
  Not Hispanic or Latino | 38 | 43 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 9 | 30
  White | 19 | 45 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 45 | 56 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Shedding for at Least One of the Influenza Strains Included in the QLAIV in the First 21 Days After Vaccine Administration Days in HIV-positive and Control Groups.
Description: Measure PCR positivity for any of the influenza subtypes included in QLAIV between baseline (day 0) and the last study visit at 14-21 days after vaccine. Compare number of participants with PCR positivity for any of the vaccine-strain influenza virus strains in each patient group.
Time Frame: 21 days
Population: HIV-infected and uninfected recipients of QLAIV; one HIV-uninfected subject was lost-to-follow-up after the first follow-up visit following vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | QLAIV, HIV-infected | QLAIV, HIV-uninfected
Number analyzed (Participants) | 45 | 56
Participants
  Baseline analysis for virus (before vaccine) | 0 | 0
  Shed any virus anytime up to 21 days post-vaccine | 30 | 28

2. Primary Outcome: Number of Participants With Shedding for at Least One of the Influenza Strains Included in the QLAIV Vaccine at Each of the 4 Study Visits, Days 0 (Baseline), 2-5, 7-10, and 14-21 in HIV-positive and Control Groups.
Description: Measure PCR positivity for any of the influenza subtypes included in QLAIV at visit 1 (day 0), visit 2 (days 2-5), visit 3 (days 7-10) and visit 4 (days 14-21). Compare number of participants with shedding for any subtype in each patient group. (The study was powered based on the 7-10 day data.)
Time Frame: day 0-21 post-vaccine
Population: Subjects with data for any of the visits
Measure: Count of Participants; unit: Participants
Arm/Group | QLAIV, HIV-infected | QLAIV, HIV-uninfected
Number analyzed (Participants) | 45 | 55
Participants
  Visit 1, day 0 | 0 | 0
  Visit 2, days 2-5: number analyzed (Participants) | 44 | 55
  Visit 2, days 2-5 | 30 | 27
  Visit 3, days 7-10: number analyzed (Participants) | 42 | 53
  Visit 3, days 7-10 | 13 | 11
  Visit 4, days 14-21: number analyzed (Participants) | 43 | 53
  Visit 4, days 14-21 | 1 | 0

3. Secondary Outcome: Number of Participants With Adverse Events Within 14 Days After Vaccination
Description: The investigators will compare the number of adverse events (AE) reported by AE category within 14 days after vaccination as reported by each participant. Data will reflect whether a participant ever reported the AE, and not the number of times the AE was reported.
Time Frame: 14 days after vaccination for AEs; up to 30 days for unscheduled visits
Measure: Count of Participants; unit: Participants
Arm/Group | QLAIV, HIV-infected | QLAIV, HIV-uninfected
Number analyzed (Participants) | 45 | 55
Participants
  Temperature >100F | 0 | 1
  Runny nose | 17 | 16
  Nasal congestion | 17 | 16
  Sore throat | 6 | 5
  Headache | 8 | 8
  Muscle aches | 8 | 2
  Decrease in energy | 11 | 3
  Decreased appetite | 6 | 2
  Any other symptom | 9 | 5
  Unscheduled medical visits in 30 days post vaccine | 2 | 10
Statistical Analysis 1: Comparison: QLAIV, HIV-infected vs QLAIV, HIV-uninfected; Test type: Equivalence — Looked for statistically-significant difference in numbers of adverse events between the two groups, used a p-value of 0.05 as the cutoff value for significance; p < 0.05, Chi-squared, Corrected; Groups were compared with Yates-corrected chi-square test or Fisher exact test for binary or categorical variables

4. Secondary Outcome: Number of Participants Reaching Seroprotection (HAI ≥ 40) Within the HIV-positive and Control Groups.
Description: The investigators will measure hemagglutinin inhibition (HAI) on blood samples #2 (14-21 days after vaccination) for all participants. The investigators will also compare the number of participants reaching HAI ≥ 40 for each virus sub-type contained in the vaccine.
Time Frame: 14-21 days
Population: The total number of participants analyzed reflect the number of subjects for whom there was a blood sample from the 4th visit at day 14-21.
Measure: Count of Participants; unit: Participants
Arm/Group | QLAIV, HIV-infected | QLAIV, HIV-uninfected
Number analyzed (Participants) | 44 | 51
Participants
  H1N1 | 35 | 35
  H3N2 | 27 | 35
  B-Victoria | 7 | 4
  B-Yamagata | 7 | 7

5. Other Pre Specified Outcome: Number of Participants With PCR-diagnosed Influenza and Clinically-diagnosed Influenza Like Illness.
Description: Compare numbers of participants with influenza diagnosed by PCR and with clinically-diagnosed influenza between the two groups. Data was taken from Influenza Infection Questionnaires #1 and #2. The last questionnaire (#2) was administered between May 15 and June 10, 2014 (after the vaccine). Data is reported as PCR-confirmed influenza and clinically-diagnosed influenza (subject told had influenza without confirmatory testing).
Time Frame: up to 11 months post-vaccination
Population: Number of participants analyzed reflects the number of subjects who participated in the end-of-season interview.
Measure: Count of Participants; unit: Participants
Arm/Group | QLAIV, HIV-infected | QLAIV, HIV-uninfected
Number analyzed (Participants) | 17 | 53
Participants
  PCR-confirmed influenza | 0 | 1
  clinically-diagnosed influenza | 2 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Description: HIV-infected and HIV-uninfected individuals
Groups:
- QLAIV, HIV-infected: Quadrivalent Live Attenuated Influenza Vaccine (QLAIV) administered to HIV-infected individuals 2 to 25 yoa
- QLAIV, HIV-uninfected: Quadrivalent Live Attenuated Influenza Vaccine (QLAIV) administered to HIV-uninfected individuals 2 to 25 yoa
Arm/Group | QLAIV, HIV-infected | QLAIV, HIV-uninfected
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/55
Other Adverse Events (participants affected / at risk) | 17/45 | 16/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QLAIV, HIV-infected (N=45) | QLAIV, HIV-uninfected (N=55)
bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — nose
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QLAIV, HIV-infected (N=45) | QLAIV, HIV-uninfected (N=55)
Temperature >100F (General disorders) | 0 (0) | 1 (1) — Temperature >100F reported at any of the 3 follow-up visits after vaccine.
Runny nose (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 16 (28) — Runny nose reported at any of the 3 follow-up visits after vaccine.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 16 (24) — Nasal congestion reported at any of the 3 follow-up visits after vaccine.
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (6) — Sore throat reported at any of the 3 follow-up visits after vaccine.
Headache (Nervous system disorders) | 8 (14) | 8 (9) — Headache reported at any of the 3 follow-up visits after vaccine.
Muscle aches (General disorders) | 8 (11) | 2 (2) — Muscle aches reported at any of the 3 follow-up visits after vaccine.
Decrease in energy (General disorders) | 11 (16) | 3 (3) — Decrease in energy reported at any of the 3 follow-up visits after vaccine.
Decreased appetite (Gastrointestinal disorders) | 6 (10) | 2 (2) — Decreased appetite reported at any of the 3 follow-up visits after vaccine.
Any other symptoms (General disorders) | 9 (9) | 5 (6) — Any other symptoms reported at any of the 3 follow-up visits after vaccine.

LIMITATIONS AND CAVEATS:
Data on influenza diagnosis from the end-of-season questionnaire is limited by the number of subjects who were available to answer the questionnaire (17/45 in HIV-infected group, 53/55 in HIV-uninfected group).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No